CLINICAL TRIAL: NCT03077932
Title: A Smartphone App to Facilitate Buprenorphine Discontinuation
Brief Title: An App to Aid in Transitioning Off Opioid Medication
Acronym: BetterOFF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 840059
Record Dates: First submitted 2017-03-08; First posted 2017-03-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Opiate Use Disorder; Opiate Withdrawal Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App Development and Open Pilot (Other): Phase 1 (app development) will consist of: 1) development of the BetterOFF prototype; and 2) series of usability studies with patients interested in discontinuing opioid medication.
  Phase 2 (open pilot) will involve conducting a 12-week open pilot trial (n=20) to test the feasibility and acceptability of the BetterOFF app with patients tapering from opiate medication.
  Interventions: Other: App Development and Open Pilot

INTERVENTIONS:
Other: App Development and Open Pilot — Phase 1 (app development) will consist of: 1) development of the BetterOFF prototype; and 2) series of usability studies with patients interested in discontinuing opioid medication.
  Phase 2 (open pilot) will involve conducting a 12-week open pilot trial (n=20) to test the feasibility and acceptability of the BetterOFF app with patients tapering from opiate medication.

SUMMARY:
The investigators propose to develop a smartphone app (called BetterOFF) that will help patients manage opioid withdrawal during opioid medication taper and detoxification. The BetterOFF smartphone intervention will be a resource patients can access anytime and anywhere. If the BetterOFF intervention were to be effective in helping patients discontinue opioid medication, it could be integrated into the standard of care of office-based clinical practices, as well as substance use programs, thereby having a substantial public health impact.

DETAILED DESCRIPTION:
Many of the growing number of patients prescribed long-term opioid medication (for a variety of reasons including a history of illicit opioid use or management of chronic pain) will express an interest in discontinuing medication. However, many patients, physically dependent on opioids, fear the withdrawal symptoms that inevitably occur with opioid medication discontinuation and will experience a decrease in their self-efficacy for abstinence at the end of a taper. As a result, tapering is often slow and done hesitantly, and relapse rates after an opioid taper are high and associated with broad consequences, including significant negative physical, mental, and social problems. Even with optimal tapering protocols, patients need novel approaches to manage the discontinuation of opiate agonist treatment. Given this important gap in opioid treatment delivery, we propose to develop a theoretically-driven, smartphone-delivered intervention (Better Off app) to help patients effectively manage the experience of opioid medication discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* between 18-65 years of age;
* currently receiving opioid medication;
* interesting in discontinuing opioid medication
* has a smartphone

Exclusion Criteria:

* non-English speaking.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Opiate use | 1 month post-taper
  Days of opiate use at follow-up

SECONDARY OUTCOMES:
Fear of withdrawal symptoms | 1 month post-taper
  Fear of withdrawal symptoms
Opiate Withdrawal | Baseline to 1 month post-taper
  opiate withdrawal symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Ana Abrantes, Ph.D., Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No